CLINICAL TRIAL: NCT05596539
Title: Prospective, Longitudinal, Observational Registry of Adult Patients With Hypophosphatasia
Brief Title: Prospective, Longitudinal, Observational Registry of Adult Patients With Hypophosphatasia (REG-HYPO)
Acronym: REG-HYPO
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220575
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Hypophosphatasia
Keywords: Cohort; Hypophosphatasia; Bone fragility; Enthesopathy; Asfotase
MeSH Terms: conditions — Hypophosphatasia; Enthesopathy | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — Collection data from diagnostic Data collected following to medical exam as part of care

SUMMARY:
The purpose of this study is to assess medical events during follow-up of adult patients having hypophosphatasia and consulting rheumatologists.

DETAILED DESCRIPTION:
Hypophosphatasia (HPP) is a rare inherited disease caused by mutations of the ALPL gene. In adult HPP, patients may suffer from fractures, pseudofractures, fracture healing complications, osteoarthritis, chondrocalcinosis, dental diseases, muscle pain and disability, but also headache, muscle weakness, ocular disease, and other symptoms. In some cases the diagnosis is severely delayed. Moreover a number of patients having such symptoms and a low level of serum alkaline phosphatase, without gene mutation can be followed by rheumatologists with difficulties in management of bone fragility and pain. The aim of this register is to describe prospectively the medical events in adult patients having hypophosphatasia, whether or not there is a proven genetic abnormality.

ELIGIBILITY:
Inclusion Criteria:

* men and women,
* aged 18 and over, with no upper age limit, who have had a total alkaline phosphatase value of less than 40 IU/l on at least 3 occasions, or at least a total alkaline phosphatase value below 40 IU/L and evidence of ALPL gene polymorphism
* with at least one rheumatological symptom.

Exclusion Criteria:

* transient hypophosphatasia: absence of confirmation of a value below 40 IU/l on at least 3 samples, lack of genetic confirmation
* secondary hypophosphatasia according to the expert rheumatologist (drugs, endocrine disease, other genetic disease...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypophosphatasia discovered in adulthood.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Characterise the circumstances of diagnosis, and deduce ways to reduce the diagnostic delay of hypophosphatasia in adults. | At inclusion
  Time since first symptom due to hypophosphatasia

SECONDARY OUTCOMES:
Characterise "non bony" forms: chondrocalcinosis, multiple tendon calcifications, inflammatory pseudo-rheumatism, odonto-HPP | At inclusion
  Proportion of each of the "non-bone" forms in the diagnosed population.
Characterise the forms for which the genetic analysis is negative | At inclusion
  Proportion of patients with clinical hypophasphatasia, without genetic evidence.
Recognise situations of associated osteoporosis. | At 72 months
  Proportion of patients with femoral and/or spinal densitometric osteoporosis.
Characterise the practical follow-up of asfotase alpha treatment started in adults | At 72 months
  Maintenance of enzyme replacement therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Christian ROUX, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (11):
- France (11):
  - CHU de Bordeaux- Hôpital Pellegrin Place Amélia Raba Léon - 12è étage - Rhumatologie -, Bordeaux, France
  - CHU Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - CHU Nice, Nice
  - Lariboisière Hospital, Paris
  - Cochin Hospital, Paris
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHU Saint-Etienne, Saint-Priest-en-Jarez
  - Les hôpitaux universitaires de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No